CLINICAL TRIAL: NCT00068848
Title: RCT of a Novel Oral Contraceptive Initiation Method
Brief Title: Quick Start Approach to Birth Control Pills
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HD42413
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2007-04-10 (Estimated); Status verified 2007-04

CONDITIONS: Pregnancy; Contraception
Keywords: Oral Contraceptives; Initiation; Continuation

INTERVENTIONS:
Behavioral: Quick start oral contraceptive initiation

SUMMARY:
Women who choose to take birth control pills are currently instructed to begin taking the pills at the end of a menstrual cycle. This creates a window of time between when the woman is given the pills and when she begins taking them. Some women fail to begin taking the pills, placing them at increased risk of pregnancy. This study will evaluate a new approach to beginning birth control pills. Women will take the first pill in the doctor's office rather than waiting until the next menstrual cycle.

DETAILED DESCRIPTION:
Despite the effectiveness of oral contraceptives, pregnancy rates are high among women who choose this method of birth control. These pregnancies occur due to incorrect use, premature discontinuation, and failure to begin taking oral contraceptives after they have been prescribed. As many as 25% of adolescents who seek oral contraceptives from family planning clinics never take the first pill. Failure to begin oral contraceptives may occur due to ambivalence, confusion about starting instructions, or intervening pregnancy. Conventional starting instructions for oral contraceptives require waiting until the next menstrual period; this may leave the woman at high risk of pregnancy. This trial will evaluate a "quick start" approach in which the woman swallows the first pill during the clinic visit under direct observation and then continues daily pill use without waiting for her next menses. The trial will determine whether immediate oral contraceptive initiation offers benefits compared to conventional starting approaches.

Participants in this study will be randomized to receive either the quick start or the standard starting approach. Participants will complete a questionnaire at study entry and Months 3 and 6. The main outcomes are 6-month oral contraceptive continuation rates and pregnancy rates.

ELIGIBILITY:
Inclusion Criteria

* Requests hormonal contraceptives as primary method of contraception
* Sexually active (intercourse within 30 days prior to study entry) or anticipating sexual activity within 30 days following study entry

Max Age: 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2000
Dates: Start 2003-02; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L. Westhoff, MD, MSc, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Emory University School of Medicine, Atlanta, Georgia
  - Mt. Sinai School of Medicine, New York, New York
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Derived] Westhoff C, Heartwell S, Edwards S, Zieman M, Cushman L, Robilotto C, Stuart G, Morroni C, Kalmuss D. Initiation of oral contraceptives using a quick start compared with a conventional start: a randomized controlled trial. Obstet Gynecol. 2007 Jun;109(6):1270-6. doi: 10.1097/01.AOG.0000264550.41242.f2. PMID 17540797